CLINICAL TRIAL: NCT01084304
Title: Assessment of Stress Levels in Consumers Using Ovulation Tests in Order to Conceive
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0172
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Stress
Keywords: Pregnancy; Ovulation tests; stress; Wishing to become pregnant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active: Use of ovulation tests to aid conception
- Control: No ovulation tests to aid conception

SUMMARY:
Approximately 150 female volunteers wishing to become pregnant will be recruited via web recruitment from around the UK and randomised 1:1 to receive Clearblue Digital ovulation tests (active arm) or no aid to conception (control arm) for 2 full menstrual cycles. All volunteers will complete study questionnaires and provide a urine sample at designated time points though out the menstrual cycle.

A sub-arm to this study, applied the same protocol to women in an infertility treatment setting; Royal Hallamshire Hospital, Sheffield. Additional exclusion criteria were applied to this cohort; had regular menstrual cycles between 25 and 35 days, and who did not have a diagnosis of bilateral or unilateral tubal blockage, documented anovulation or severe male-factor infertility (with <5 million motile sperm per ejaculate). For this arm, the protocol was reviewed by Sheffield Research Ethics Committee 09/H1308/134.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study and agree to comply with study procedures.
* Has menstrual bleeds.
* Seeking to become pregnant.
* Living in UK

Exclusion Criteria:

* Used hormonal contraception within the last 3 months.
* Currently undergoing fertility treatment or investigation.
* Diagnosed as infertile following investigations.
* Drug or alcohol dependency.
* history of depression, anxiety or panic attacks

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females aged 18 to 40 wishing to become pregnant
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cortisol Measurement | Twice monthly
  Measurement of Urinary Cortisol throughout menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Dr, Principal Investigator
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

REFERENCES:
- [Derived] Jones G, Carlton J, Weddell S, Johnson S, Ledger WL. Women's experiences of ovulation testing: a qualitative analysis. Reprod Health. 2015 Dec 21;12:116. doi: 10.1186/s12978-015-0103-y. PMID 26689590
- [Derived] Tiplady S, Jones G, Campbell M, Johnson S, Ledger W. Home ovulation tests and stress in women trying to conceive: a randomized controlled trial. Hum Reprod. 2013 Jan;28(1):138-51. doi: 10.1093/humrep/des372. Epub 2012 Oct 18. PMID 23081872